CLINICAL TRIAL: NCT04341337
Title: Evaluation of Ethical Implication of a Training Model Necessary to Gain Access to a Surgical Innovation Device.
Brief Title: Link of Interest and Training Model
Status: Completed | Type: Observational
Sponsor: Centre de l'arthrose, Paris (Other)
Responsible Party: Principal Investigator, Maillot Cédric, principal investigator, Centre de l'arthrose, Paris
Other Study IDs: pipac
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- expert: interviews of expert of pipac about ethical issues
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — questionnaire about ethics in surgery

SUMMARY:
* The surgical device used to perform PIPAC procedure is commercialized by a single manufacturer under a monopoly regimen, and a formal training (economically supported by the manufacturer) is mandatory for surgeons who want to buy the device.Relations with the company and solutions to extend training require specific analysis from an ethical point of view.
* Based on the growing number of published papers from a growing number of international centers, the controlled training model is not limiting, and it is a successful model of development of this breakthrough innovation.
* But with the major involvement of the industry and the control of training, the different levels of interest could induce ethical questions.

DETAILED DESCRIPTION:
* Objective: Using the example of Pressurized Intra Peritoneal Aerosol Chemotherapy (PIPAC), the investigators analyze the development model of this procedure and provide an ethical analysis of the involvement of the industry in this development.
* Summary Background Data: In the case of breakthrough innovation, medical training is essential for safe use of the new procedure. Pharmaceutical companies may organize this training; but when it becomes the only training opportunity to use the device, scientists and clinicians are exposed to a conflict of interest.
* Methods: The investigators performed a literature review of PIPAC publications using the STROBE criteria. Then, the investigators conducted interviews with an expert panel to analyze the ethical impact of involvement of the industry in the development of the PIPAC procedure.

ELIGIBILITY:
Inclusion Criteria:

* expert in pipac
* more than 30 PIPAC per year

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: expert working in academic tertiary center
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
qualitative analysis of the interviews | 1 month
  Questions for interviews were first prepared. Six questions for the clinicians and the scientist were elaborated about the interviewees' experience concerning the initiation and use of PIPAC, difficulties encountered to initiate this activity in their respective centres, description of the involvement of the industry for the development of the technique, the clinician-industry relationship, the mandatory nature of the training, and their ethical judgment on this model. For the biomedical manager, questions were about the set-up of the PIPAC procedure and the implication of the industry in the process. The commercial representative was interviewed about the business strategy of the industry. The interviewer had the freedom to adapt questions to prior answers. Interviewees did not receive the questionnaire before the discussion.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martellotto S, Maillot C, Villeneuve L, Eveno C, Sgarbura O, Pocard M. Restricted access to innovative surgical technique related to a specific training, is it ethical? Example of the PIPAC procedure. A systematic review and an experts survey. Int J Surg. 2020 Nov;83:235-245. doi: 10.1016/j.ijsu.2020.07.004. Epub 2020 Jul 29. PMID 32738543